CLINICAL TRIAL: NCT01863927
Title: The Effect of Ventilated Vest on Thermoregulation During Exercise in Hot
Brief Title: The Effect of Ventilated Vest on Thermoregulation During Exercise in Hot Environment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Barliz Adato, Head Physician at the Institute of Military Physiology, Heller Institute of Medical Research, Sheba Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SHEBA-12-9726-AD-CTIL; 1178-12 (Other: IDF)
Record Dates: First submitted 2013-05-23; First posted 2013-05-29 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Body Temperature Changes
MeSH Terms: conditions — Body Temperature Changes | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Research arm (Experimental): Each of the participants will be randomly exposed to 4 conditions during four separate consecutive days.
  Interventions: Other: Research intervention

INTERVENTIONS:
Other: Research intervention — After heat acclimation the participant will be randomly exposed to 4 conditions during four separate consecutive days: 1) walking on a treadmill for two hours in hot-wet conditions (30OC, 70% RH) while wearing military uniforms and a vest (control group); 2) walking on a treadmill for two hours in hot-dry conditions (40OC, 30% RH) while wearing military uniforms and a vest (control group); 3) walking on a treadmill for two hours in hot-wet conditions (30OC, 70% RH) while wearing military uniforms and a vest with a ventilator (experimental group); 4) walking on a treadmill for two hours in hot-dry conditions (40OC, 30% RH) while wearing military uniforms and a vest with a ventilator (experimental group)
  Other Names: Heat exposure, exercise in hot environment

SUMMARY:
The purpose of this preliminary experiment is to measure the effect of a novel ventilation system on the physiological strain during exercise in high heat load while wearing ballistic protective vest. Ten young and healthy participants will participate in the study. They will all go through a six days heat acclimation period in a heat chamber according to a valid protocol. Afterwards they will be randomly exposed to 4 conditions during four separate consecutive days.

DETAILED DESCRIPTION:
Ten young and healthy civilian participants will participate in the study. They will all go through a six days heat acclimation period in a heat chamber according to a valid protocol. After heat acclimation the participant will be randomly exposed to 4 conditions during four separate consecutive days: 1) walking on a treadmill for two hours in hot-wet conditions (30OC, 70% RH) while wearing military uniforms and a vest (control group); 2) walking on a treadmill for two hours in hot-dry conditions (40OC, 30% RH) while wearing military uniforms and a vest (control group); 3) walking on a treadmill for two hours in hot-wet conditions (30OC, 70% RH) while wearing military uniforms and a vest with a ventilator (experimental group); 4) walking on a treadmill for two hours in hot-dry conditions (40OC, 30% RH) while wearing military uniforms and a vest with a ventilator (experimental group). During the heat exposures, rectal temperature, skin temperature and heart rate will be continuously monitored. Subjective comfort measures, heat strain indices, sweat rate and sweat evaporation will be also measured/calculated. The differences in the above measures, during exposure to exercise in the heat between ventilator and no ventilator will be then analyzed.

ELIGIBILITY:
Inclusion Criteria:

* age 21-28
* healthy
* after medical checkup
* after signing concent form

Exclusion Criteria:

* heart disease
* respiratory disease
* baseline bp above 140/90 mmHg
* sleep disorders
* diabetes
* anhydrosis
* skin disease
* acute illness in last 3 days prior to the examination

Ages: 21 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-11 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Heat tolerance test | 1 year
  The test is performed in a climatic chamber at a temperature of 40oC and 40% relative humidity. During the test, the subject walks on a treadmill at a speed of 5 km/hr at a 2% grade for 2h. Body core temperature and heart rate are continuously monitored, and sweat rate is computed from body weight prior to and after the test, corrected for fluid intake. Heat intolerance is determined when body core temperature elevates above 38.5oC, when heart rate elevates above 150 bpm, or when either does not tend to reach a plateau.
Maximal oxygen consumption test | 1 year
  Volunteer's oxygen consumption (VO2) will be monitored continuously with a metabolic chart (ZAN), while running for 10 min on a treadmill under comfortable environmental conditions.

SECONDARY OUTCOMES:
Skin temperature | 1 year
  The volunteers will undergo heat tolerance test. Their skin temperature will be measured by skin thermistors and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Rectal temperature | 1 year
  The volunteers will undergo heat tolerance test. Their rectal temperature will be measured by rectal thermistor and will be monitored continuously and viewed by the attending medical staff. Automatically all data will be recorded by the monitoring Biopac system.
Heart rate | 1 year
  During the HTT and the VO2 test heart rates will be monitored continuously and will be stored by a heart rate wristwatch, (POLAR, Finland).

CONTACTS AND LOCATIONS:
Overall Officials: Barliz Adato, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba medical center, Tel-Hashomer, Ramat- Gan, Israel